CLINICAL TRIAL: NCT04332471
Title: Treatment of Plantar Fasciitis With Radial Shockwave Therapy vs. Focused Shockwave Therapy: a Randomized Controlled Trial
Brief Title: Shockwave Therapy for Plantar Fasciitis RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-1517
Record Dates: First submitted 2020-03-11; First posted 2020-04-02 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Plantar Fascitis
MeSH Terms: interventions — Home Infusion Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Control (Active Comparator): Patients in the control group will be treated using the home therapy protocol only.
  Interventions: Other: Home therapy
- Radial shockwave therapy (Active Comparator): Patients will receive 4 sessions of radial shockwave therapy.
  Interventions: Procedure: Radial shockwave therapy; Device: Shockwave therapy device; Other: Home therapy
- Focused shockwave therapy (Active Comparator): Patients will receive 4 sessions of focused shockwave therapy.
  Interventions: Procedure: Focused shockwave therapy; Device: Shockwave therapy device; Other: Home therapy

INTERVENTIONS:
Procedure: Radial shockwave therapy — Target intensity will be within a range of 3.5-5.0 bar at maximum Hz, titrated up to patient tolerance within 100 pulses. Total of 3000 pulses.
  Arms: Radial shockwave therapy
Procedure: Focused shockwave therapy — Target intensity will be within a range of 0.15-0.25 mJ/mm2 at maximum Hz, titrated up to patient tolerance within 100 pulses. Total of 3000 pulses.
  Arms: Focused shockwave therapy
Device: Shockwave therapy device — The shockwave therapy device will be used to administer either radial or focused shockwave therapy.
  Arms: Focused shockwave therapy; Radial shockwave therapy
Other: Home therapy — Stretching and ice massage

SUMMARY:
Inflammation of the plantar fascia is known as plantar fasciitis and is commonly seen in active or overweight individuals. It can be treated via conservative or surgical therapies. Extracorporeal shockwave therapy has shown promise in the treatment of plantar fasciitis. Several studies have compared the effects of different types of extracorporeal shockwave therapy (radial and focused) with other forms of conservative treatment in patients with chronic plantar fasciitis. No study has yet compared the effect of radial vs. focused shockwave therapy on pain in this population.

DETAILED DESCRIPTION:
Plantar fasciitis is a common foot problem that affects 3.8 per 1,000 persons in the United States. It is characterized by inflammation of the plantar fascia, a fibrous tissue which connects the calcaneus to the metatarsal heads, and is often seen in individuals who are overweight and/or participate frequently in weight-bearing endurance activities such as running. Pain is typically at its highest during the first steps in the morning, although it can also occur with prolonged weightbearing. Plantar fasciitis can be treated via conservative or surgical measures, although surgery is considered as the last resort. In recent years, extracorporeal shockwave therapy has emerged as an alternative conservative method for treating plantar fasciitis. There are two types -- radial and focused shockwave therapy. Focused therapy creates deeper-penetrating, higher-energy shockwaves, whereas radial therapy produces more superficial shockwaves that can treat a wider area of pathology.

Randomized controlled trials have compared focused and radial shockwave therapy to placebo and other conservative measures in the treatment of chronic plantar fasciitis and overall demonstrated benefit. Only one study has directly compared radial and focused shockwave therapy in this population, although pain was not an outcome of focus in the study. The current study aims to collect patient-reported outcomes on both pain and function following radial vs. focused shockwave therapy vs. control therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with a clinical diagnosis of chronic plantar fasciitis (>3 months) that has been recalcitrant to other treatments
* Minimum VAS pain of 40/100 (4/10; morning pain when taking first steps, pain after prolonged walking/standing)
* English-speaking

Exclusion Criteria:

* Cortisone injection within the past 3 months
* Platelet-rich plasma injection within the past 6 months
* History of previous foot surgery
* Bilateral heel pain
* Coagulopathies or use of anti-coagulants
* Local and systemic neurologic or vascular insufficiencies
* Rheumatologic disorders
* Systemic inflammatory disorders
* Active or chronic infection in the area
* Lower extremity bone disorders (e.g., Paget's disease, osteomyelitis)
* Calcaneal fractures
* Nerve entrapment
* Ruptures in tendon
* Non-English speaking

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale pain - morning | Up to 1 year
  Morning pain. This will be assessed on a scale of 0-100, with a higher score representing more pain.
Visual analog scale pain - after prolonged walking or standing | Up to 1 year
  Pain after prolonged walking or standing. This will be assessed on a scale of 0-100, with a higher score representing more pain.

SECONDARY OUTCOMES:
PROMIS Physical Function computer adaptive test score | Up to 1 year
  This computer adaptive questionnaire assesses physical function. A higher score represents higher function. A score of 50 represents the population average.
Foot and Ankle Outcome Score (FAOS) | Up to 1 year
  The FAOS assess pain, symptoms, activities of daily living, sports, and quality of life related to foot and ankle pain. This will be assessed on a scale of 0-100, where 100 indicates no problems and 0 indicates extreme problems.
Treatment satisfaction | Up to 1 year
  Satisfaction with the assigned treatment will be determined on a 0-10 scale, with 10 being most satisfied and 0 being least satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Quirolgico, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States